CLINICAL TRIAL: NCT06485973
Title: Evaluation of Dental Anxiety in Patients Undergoing Different Dental Treatments - A Prospective Study
Brief Title: Dental Anxiety in During Different Dental Treatments (DENANX)
Acronym: DENANX
Status: Completed | Type: Observational
Sponsor: Asst. Prof. Dr. Suleyman Emre Meseli (Other)
Responsible Party: Sponsor-Investigator, Asst. Prof. Dr. Suleyman Emre Meseli, Assoc. Prof. Suleyman Emre MESELI, PhD, DDS, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Other Study IDs: IAUDENT-01
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants who are involved in the treatment planning of any of the following treatments: filling, root canal treatment, scaling, implant treatment and tooth extraction.
  Interventions: Other: Modified Dental Anxiety Scale (MDAS)

INTERVENTIONS:
Other: Modified Dental Anxiety Scale (MDAS) — The MDAS is described as a scale to provide a more comprehensive assessment of dental anxiety. The MDAS has shown favorable psychometric properties with acceptable reliability and validity.

SUMMARY:
The aim of this observational cross-sectional study is to evaluate the dental anxiety levels of participants aged 18-70 years who will scheduled for different dental treatmentsThe main question it aims to answer is:

Does the type of dental treatment make a difference in the level of dental anxiety in participants? Within the scope of their dental treatment, participants who have already been planned to assign any of the filling, root canal treatments, scaling, tooth extraction and implant placement will have their anxiety levels recorded through a questionnaire just before starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation
* sufficient Turkish literacy
* no recent psychiatric diagnoses within the previous year
* no psychotherapy in the past six months,
* and no use of psychotropic drugs or illicit substances that could affect mental health in the previous year.

Exclusion Criteria:

-To stop volunteering until the study is completed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cross-sectional survey-based research will be conducted on 322 volunteers aged 18 to 70 at Istanbul Aydin University Faculty of Dentistry between March 1, 2021, and April 30, 2021. Participants will be included in the study if they met the following criteria: voluntary participation, sufficient Turkish literacy, no recent psychiatric diagnoses within the previous year, no psychotherapy in the past six months, and no use of psychotropic drugs or illicit substances that could affect mental health in the previous year.
  After a comprehensive oral and dental examination, an individualized treatment plan will be developed for each participants. These plans includes necessary dental procedures, such as fillings, root canals, scaling, tooth extractions, and implant procedures. The participants will be scheduled to receive their treatments on the seventh day, according to their individual needs. On that day, they will complete a survey while waiting in the waiting room.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Dental Anxiety Scale | 1 hour
  The data collection tool is an 8-question, 4-point Likert-type scale based on the MDAS, which has been validated for reliability and accuracy. The questions is designed to assess the anxiety levels of participants prior to scheduled dental procedures.
  The participants' responses are scored on a scale of 0-3 to indicate their level of anxiety and stress. A score of 0 indicated no anxiety, 1 indicated mild anxiety, 2 moderate indicated anxiety, and 3 indicated severe anxiety and stress. The dental anxiety level is determined based on the sum of scores given to the eight relevant questions, which ranged from 0 to 24 and is used to calculate the MDAS score. The MDAS score is then compared to the following cut-off values to determine the level of dental anxiety: a score of 0 indicated no anxiety, 1-8 indicated mild anxiety, 9-16 indicated moderate anxiety, and 17-24 indicated severe anxiety.

SECONDARY OUTCOMES:
Demographical Outcomes | 1 hour
  Demographic outcomes are as follows; age, sex, marital status, number of children, education level, and occupation.
Oral and Dental Health Experiences and Attitudes | 1 hour
  To assess participants' experiences and attitudes toward oral and dental health, including frequency of toothbrushing and dental treatment, previous dental experiences, and pre-treatment anxiety levels. In the questionnaire, which is a data collection tool, the frequency of tooth brushing is asked with the options of 1/day / 2 times a day / 1/week / 2-3 times a week, and the dental treatments in the past are asked to mark. They were also asked to tick how they found their experience (good/medium/bad) following these treatments. There are multiple choice questions to understand the presence of dental anxiety before treatment and what triggers it.
Dental Anxiety Assessment | 1hour
  To assess participants' experience of dental anxiety, including its level, cause, onset, physical symptoms, and coping mechanisms. Additionally, it will be examined environmental triggers that contribute to dental anxiety, such as noise from equipment and the sight of sharp instruments, and the length of time it took for anxiety to peak. The objective of this section is to provide a comprehensive understanding of the participants' dental anxiety, its causes, and their self-coping strategies, as well as the impact of environmental factors on their anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appukuttan DP. Strategies to manage patients with dental anxiety and dental phobia: literature review. Clin Cosmet Investig Dent. 2016 Mar 10;8:35-50. doi: 10.2147/CCIDE.S63626. eCollection 2016. PMID 27022303
- [Background] Humphris G, Crawford JR, Hill K, Gilbert A, Freeman R. UK population norms for the modified dental anxiety scale with percentile calculator: adult dental health survey 2009 results. BMC Oral Health. 2013 Jun 24;13:29. doi: 10.1186/1472-6831-13-29. PMID 23799962
- [Result] Kassem El Hajj H, Fares Y, Abou-Abbas L. Assessment of dental anxiety and dental phobia among adults in Lebanon. BMC Oral Health. 2021 Feb 4;21(1):48. doi: 10.1186/s12903-021-01409-2. PMID 33541354